CLINICAL TRIAL: NCT03495154
Title: A Multi-center Post-market Single Arm Prospective Study of Parietene™ DS Composite Mesh in Subjects Undergoing Ventral Hernia Repair
Brief Title: Post Market Study of Parietene™ DS Composite Mesh in Ventral Hernia Repair
Acronym: PPDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17051PDS
Record Dates: First submitted 2018-03-27; First posted 2018-04-11 (Actual); Results first posted 2022-11-17 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Masking Description: All subjects enrolled will receive the Parietene DS Composite Mesh
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Parietene DS Composite Mesh (Experimental): Patients treated with Parietene DS Composite Mesh
  Interventions: Device: Parietene DS Composite Mesh

INTERVENTIONS:
Device: Parietene DS Composite Mesh — All subjects enrolled will receive the Parietene DS Composite Mesh

SUMMARY:
A multi-center post-market single arm prospective study of Parietene™ DS Composite Mesh in subjects undergoing ventral hernia repair to confirm its clinical safety and performance in the short (1, 3 months), mid (12 months) and long term (24 months)

DETAILED DESCRIPTION:
A multi-center post-market single arm prospective study of Parietene™ DS Composite Mesh in subjects undergoing ventral hernia repair to confirm its clinical safety and performance in the short (1, 3 months), mid (12 months) and long term (24 months)

125 male or female adults subjects will be enrolled in a minimum of 4 USA sites who are undergoing elective ventral hernia repair (primary or incisional)

ELIGIBILITY:
Inclusion Criteria:

* Preoperative Inclusion Criteria

  1. Subject has provided informed consent
  2. Subject is ≥18 years of age (at the time of consent)
  3. Subject is undergoing elective ventral hernia repair (primary or incisional) with intraperitoneal mesh placement

Exclusion Criteria:

* Preoperative Exclusion Criteria

  1. BMI > 45 kg/m2
  2. Subject is undergoing emergency surgery
  3. Subject is pregnant or planning to become pregnant during study participation period
  4. Subject is unable or unwilling to comply with the study requirements or follow-up schedule
  5. Subject has comorbidities which, in the opinion of the Investigator, will not be appropriate for the study or the subject has an estimated life expectancy of less than 6 months
  6. The subject has participated in another investigational drug or device research study within 30 days of enrollment
  7. Subject has a parastomal hernia
* Intra-operative Exclusion Criteria

  1. Subject's hernia repair is in a contaminated or infected site (CDC wound class 2-4) as assessed by the Investigator(s)
  2. Subject is undergoing "bridging" repair technique with the mesh placed in an "inlay" position
  3. Surgeon is unable to completely remove existing mesh from prior surgery
  4. Surgeon overlays 2 meshes
  5. Subject receives any mesh other than Parietene™ DS composite mesh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Kim, Study Director — Medtronic - Surgical Innovations
Locations (6):
- United States (6):
  - Our Lady of the Lakes Regional Medical Center, Baton Rouge, Louisiana
  - University of Missouri - Columbia, Columbia, Missouri
  - The Ohio State University, Columbus, Ohio
  - Hernia Center of Excellence LLC, Newport News, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parietene DS Composite Mesh
Started | 145 (There were 145 subjects screened and consented.)
Full Analysis Set | 125 (Full Analysis Set (FAS) includes any enrolled subject who received study device. Results are based on Full Analysis Set subjects.)
Completed | 104 (Number of subjects that completed the study)
Not Completed | 41
Not completed — Screen Failures Pre-Operatively | 4
Not completed — Withdrawn Prior to Surgery | 10
Not completed — Screen Failures During Surgery | 6
Not completed — Death | 2
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 2
Not completed — Unable to gather information from subject due to age and limited abilities | 1

BASELINE CHARACTERISTICS:
Population: Post Market Study of Parietene™ DS Composite Mesh in Ventral Hernia Repair
  Approximately 125 Subjects
Arm/Group | Parietene DS Composite Mesh
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years]
  Overall | 58.0 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 125
Ethnicity [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 22
  White | 98
  Latino/Hispanic | 2
  Middle Eastern | 1
  Patient Does Not Want to Disclose | 1
Height, cm [Mean (Standard Deviation); unit: centimeters] | 172.5 (11.15)
Weight, kg [Mean (Standard Deviation); unit: kilograms] | 98.4 (15.96)
BMI, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 33.2 (4.82)
Pregnancy Test Performed [Count of Participants; unit: Participants] — Population: [1] Measure Analysis Population Description: Pregnancy test was only performed for female subjects of child bearing age and potential. Pregnancy tests for women are request at the time of screening and operation except for women who are post-menopausal for at least 2 years or surgically sterile. If screening was done the same day of operation (as permitted by CIP), only one pregnancy test is necessary.
  Participants
    Pregnancy Test at Screening Visit: number analyzed (Participants) | 51
    Pregnancy Test at Screening Visit: Pregnancy Test Administered: Yes | 10
    Pregnancy Test at Screening Visit: Pregnancy Test Administered: No | 41
    Pregnancy Test at Operative Visit: number analyzed (Participants) | 27
    Pregnancy Test at Operative Visit: Pregnancy Test Administered: Yes | 5
    Pregnancy Test at Operative Visit: Pregnancy Test Administered: No | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hernia Recurrence Within 12 Months Following Parietene™ DS Composite Mesh Use in Ventral Hernia Repair
Time Frame: 12 months post surgery
Population: Hernia recurrence rate at 12M changed from what was previously reported, 4 (3.5%) due to data imputed for hernia recurrence. It was assumed subjects who missed the 12M visit and had no recurrence at 24M also had no recurrence at 12M, as hernias cannot appear and then disappear over time without treatment. There were 5 subjects excluded from the primary endpoint analysis due to not completing the 12M/24M visits and therefore, unable to determine if a recurrence occurred in these subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Parietene DS Composite Mesh
Number analyzed (Participants) | 120
Participants
  Subjects With Hernia Recurrence at 12-Months | 4
  Subjects Without Hernia Recurrence at 12-Months | 116
Statistical Analysis 1: Comparison: Parietene DS Composite Mesh; Number of participants with hernia recurrence within 12 months following Parietene™ DS Composite Mesh use in ventral hernia repair; Test type: Other — This was not a comparative endpoint; Percentage and confidence interval = 3.3, 95% CI 2-sided [1.0 to 8.5]

2. Secondary Outcome: Number of Participants With Incidence of Adverse Device Effects (ADEs) Intra-operatively, at Discharge, Within 1 Month, 3 Months, 12 Months and 24 Months Following Parietene™ DS Composite Mesh Use in Ventral Hernia Repair.
Time Frame: operation, discharge, 1 month, 3 months, 12 months and 24 months post surgery
Measure: Number; unit: number of participants with ADEs
Arm/Group | Parietene DS Composite Mesh
Number analyzed (Participants) | 125
number of participants with ADEs
  Number of participants with incidence of ADEs Intra-Operatively | 0
  Number of participants with incidence of ADEs at Discharge | 14
  Number of participants with incidence of ADEs within 1 Month | 31
  Number of participants with incidence of ADEs within 3 Months | 34
  Number of participants with incidence of ADEs within 12 Months | 40
  Number of participants with incidence of ADEs within 24 Months | 42
Statistical Analysis 1: Comparison: Parietene DS Composite Mesh; Test type: Other — Statistical Analysis is based on number of participants with incidence of with ADEs at discharge. Adverse Device Effects (ADE) is inclusive of both procedure and/or device related AEs; Number of Subjects with ADEs = 14
Statistical Analysis 2: Comparison: Parietene DS Composite Mesh; Test type: Other — Statistical Analysis is based on number of participants with incidence of ADEs within 1 month. Adverse Device Effects (ADE) is inclusive of both procedure and/or device related AEs; Number of Subjects with ADEs = 31
Statistical Analysis 3: Comparison: Parietene DS Composite Mesh; Test type: Other — Statistical Analysis is based on number of participants with incidence of ADEs within 3 months. Adverse Device Effects (ADE) is inclusive of both procedure and/or device related AEs; Number of Subjects with ADEs = 34
Statistical Analysis 4: Comparison: Parietene DS Composite Mesh; Test type: Other — Statistical Analysis is based on number of participants with incidence of ADEs within 12 months. Adverse Device Effects (ADE) is inclusive of both procedure and/or device related AEs; Number of Subjects with ADEs = 40
Statistical Analysis 5: Comparison: Parietene DS Composite Mesh; Test type: Other — Statistical Analysis is based on number of participants with incidence of ADEs within 24 months. Adverse Device Effects (ADEs) are inclusive of both procedure and device related AEs; Number of Subjects with ADEs = 42

3. Secondary Outcome: Number of Participants With Incidence of Hernia Recurrence at 1 Month, 3 Months and 24 Months Following Parietene™ DS Composite Mesh Use in Ventral Hernia Repair
Time Frame: 1 month, 3 months, and 24 months post-surgery
Population: The overall number of participants analyzed may vary at different follow-up time points due to some assessments not being completed, which are required for inclusion in the analysis. At Baseline and Procedure there were 125 patients treated; each follow-up visit was missing some of those treated patients. Pre-specified full analysis set was inclusive of patients that missed follow-up. Subjects were not considered lost to follow-up until the 24M follow-up period was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Parietene DS Composite Mesh
Number analyzed (Participants) | 125
Participants
  Participants with hernia recurrence within 1 month: number analyzed (Participants) | 124
  Participants with hernia recurrence within 1 month | 0
  Participants with hernia recurrence within 3 months: number analyzed (Participants) | 123
  Participants with hernia recurrence within 3 months | 0
  Participants with hernia recurrence within 24 months: number analyzed (Participants) | 106
  Participants with hernia recurrence within 24 months | 4
Statistical Analysis 1: Comparison: Parietene DS Composite Mesh; Test type: Other — This was not a comparative endpoint; % of Subjects with Recurrence within 1M = 0, 95% CI 2-sided [0 to 2.9]
Statistical Analysis 2: Comparison: Parietene DS Composite Mesh; Test type: Other — This was not a comparative endpoint; % of Subjects with Recurrence within 3M = 0, 95% CI 2-sided [0 to 3.0]
Statistical Analysis 3: Comparison: Parietene DS Composite Mesh; Test type: Other — This was not a comparative endpoint; % of Subjects with Recurrence within 24M = 4, 95% CI 2-sided [1.2 to 9.6]

ADVERSE EVENTS:
Time Frame: Starting at the time the participant is enrolled and receives the study device up to and including 24 months post-operative
Description: Adverse events (AE) is defined in the PPDS protocol as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. Serious adverse event (SAE) definition in PPDS protocol is consistent with definition defined by clinicaltrials.gov.
Arm/Group | Parietene DS Composite Mesh
All-Cause Mortality (participants affected / at risk) | 2/125
Serious Adverse Events (participants affected / at risk) | 29/125
Other Adverse Events (participants affected / at risk) | 20/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parietene DS Composite Mesh (N=125)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
Abdominal Wall Abscess (Infections and infestations) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
COVID-19 Pneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Hemoglobin Decreased (Investigations) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuroendocrine Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Breast Necrosis (Reproductive system and breast disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pacemaker Generated Rhythm (Surgical and medical procedures) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Ileus (General disorders) | 3 (3)
Internal Hernia (Gastrointestinal disorders) | 1 (1)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parietene DS Composite Mesh (N=125)
Seroma (Injury, poisoning and procedural complications) | 13 (13)
Abdominal Pain (Gastrointestinal disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03495154/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03495154/SAP_001.pdf